CLINICAL TRIAL: NCT06167837
Title: Efficacy of Metoclopramide for Gastric Visualization by Endoscopy in Patients With Active Upper Gastrointestinal Bleeding: Multicenter, Double-blind Randomized Controlled Trial
Brief Title: Metoclopramide for Gastric Visualization in Active Upper GI Bleeding
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: King Chulalongkorn Memorial Hospital (Other)
Responsible Party: Principal Investigator, Rapat Pittayanon, Associate Professor, King Chulalongkorn Memorial Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Metoclopramide.UGIB
Record Dates: First submitted 2023-09-30; First posted 2023-12-13 (Actual); Last update posted 2023-12-13 (Actual); Status verified 2023-12

CONDITIONS: Upper GI Bleeding
Keywords: active upper GI bleeding; EGD; Gastric visualization; Metoclopramide
MeSH Terms: conditions — Gastrointestinal Hemorrhage | interventions — metoclopramide sulfone; Saline Solution; Injections

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Metoclopramide group (Experimental): Metoclopramide 10 mg +NSS 10ml IV 30-60 min before EGD
  Interventions: Drug: Metoclopramide Sulfone
- Placebo group (Placebo Comparator): NSS 10 ml IV 30-60 min before EGD
  Interventions: Drug: Normal Saline 10 mL Injection

INTERVENTIONS:
Drug: Metoclopramide Sulfone — Metoclopramide 10mg+NSS 10 ml IV 30-60 minutes before EGD
  Arms: Metoclopramide group
Drug: Normal Saline 10 mL Injection — Normal saline 10 ml IV 30-60 minutes before EGD
  Arms: Placebo group

SUMMARY:
This study aim to evaluate the efficacy of metoclopramide for gastric visualization in patients with active UGIB. This is a double-blinded, multicenter RCT. Patients with 'active' UGIB (hematemesis or presence of fresh blood in the nasogastric tube) were enrolled. The eligible patients were randomly assigned in a concealed 1:1 allocation to received either intravenous metoclopramide or placebo before endoscopy. The primary outcome was 'adequate visualization' by objective endoscopic visualized scores(EVS). Secondary outcomes included mean difference in total EVS and EVS at each location , duration of EGD, immediate hemostasis, need for a second look EGD, units of blood transfusion, length of hospital stay and 30-day rebleeding rate.

DETAILED DESCRIPTION:
* This is double-blinded, multicenter RCT including six hospitals in Thailand.
* The participated endoscopists had work experience for endoscopy more than three years.
* All endoscopists at six participating sites attended the pre-study meeting for standardization of the protocol and scoring system.
* The primary outcome was 'adequate visualization' by objective endoscopic visualized scores(EVS). ; To assess overall endoscopic visualization, we estimated the coverage of a blood clot on mucosa in four locations including 1) gastric fundus, 2) corpus, 3) antrum and 4) duodenal bulb, according to the reference endoscopic views in protocal.
* All photos, including the reference endoscopic views, were taken and internally validated by another endoscopist who was blinded to the randomization allocation.
* This study includes pre-specified subgroup analysis by location of bleeding including gastric subgroup analysis.

ELIGIBILITY:
Inclusion Criteria:

* All adult patients (aged ≥ 18years)
* Active UGIB who arrived at emergency room (ER) and had a schedule for EGD within 12 hours after onset of bleeding ; Active UGIB was defined as having hematemesis or fresh blood by diagnostic gastric lavage at the ER.

Exclusion Criteria:

* known allergy to metoclopramide
* prior gastric or duodenal surgery
* known case of esophageal, gastric or duodenal cancer;
* advanced HIV infection (defined as WHO criteria13-15: CD4 <200 cell/mm3 or WHO clinical stage 3 or 4)
* pregnancy
* gastric lavage was performed with solution > 50 ml.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 220 (Estimated)
Dates: Start 2023-10-01 (Actual); Primary Completion 2025-05-01 (Estimated); Study Completion 2025-06-30 (Estimated)

PRIMARY OUTCOMES:
Percentage of patients with 'adequate visualization' | Through study completion, estimate 2 years
  'adequate visualization' is determined by objective scoring method (endoscopic visualized scores (EVS) to estimate the coverage of a blood clot on mucosa in four locations including 1) gastric fundus, 2) corpus, 3) antrum and 4) duodenal bulb; At each location was assessed and scored between 0 and 2: 0, blood clot cover more than 75% of the surface ; 1, 25-75% blood clot coverage ; 2, blood clot coverage less than 25%. ; score >=6 considered as adequate visualization

SECONDARY OUTCOMES:
The mean difference in EVS | Through study completion, estimate 2 years
  total of four locations and at each location including fundus, corpus, antrum and duodenal bulb
Duration of esophagogastroduodenoscopy | 10minutes to 2 hours
Immediate hemostasis | Through study completion, estimate 2 years
  Rate of succession of hemostasis (bleeding stop) at first EGD
The need for a second look EGD within 72 hours after initial endoscopy | Up to 72 hours
  Rate of need for a second look EGD within 72 hours after initial endoscopy The 72-hour recurrent GI bleeding was documented and re-EGD was performed to confirm rebleeding if the following conditions were met: I) hematemesis or bloody nasogastric tube (NG) > 6 hours after endoscopy; II) melena after normalization of stool color; III) hematochezia after normalization of stool color or melena; IV) development of tachycardia (HR ≥ 110 bpm) or hypotension(SBP ≤ 90 mmHg) after ≥ 1 hour of vital sign stability without other cause; V) hemoglobin drop of ≥ 2 g/dL after two consecutive stable hemoglobin values ( < 0.5 g/dL decrease) ≥ 3 hours apart; VI) tachycardia or hypotension that does not resolve within 8 hours after index endoscopy despite appropriate resuscitation (in the absence of an alternative explanation), associated with persistent melena or hematochezia or; VII) persistently dropping hemoglobin of > 3 g/dL in 24 hours associated with persistent melena or hematochezia.
Number of unit of red blood cell transfusion during first 24 hours | Up to 24 hours
  Number of of unit of red blood cell transfusions during first 24 hours
Length of hospital stays | 1day - 30days
  Length of hospital stays of participants
30-day rebleeding rate | Up to 30 days
  rate of 30-day rebleeding of upper GI tract

CONTACTS AND LOCATIONS:
Locations (2):
- Thailand (2):
  - King Chulalongkorn memorial hospital, Bangkok
  - King Chulalongkorn Memorial hospital, Bangkok

IPD SHARING:
Plan to Share IPD: No